CLINICAL TRIAL: NCT02537262
Title: Effect of Preoperative Oral Carbohydrates on Quality of Recovery in Laparoscopic Colorectal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2015-0451
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Disease
Keywords: carbohydrate; quality of recovery(QOR) 40; enhanced recovery after surgery(ERAS)

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- carbohydrate group (Experimental)
  Interventions: Dietary Supplement: carbohydrate beverage
- NPO(None Per Oral) group (Placebo Comparator)
  Interventions: Dietary Supplement: NPO(None Per Oral)

INTERVENTIONS:
Dietary Supplement: carbohydrate beverage — Carbohydrate group drinks carbohydrate beverage 400ml(9PM~MN) the day before the surgery and 200ml three hours before the surgery.
  Arms: carbohydrate group
Dietary Supplement: NPO(None Per Oral) — NPO group does not drink any water from the MN before the surgery.
  Arms: NPO(None Per Oral) group

SUMMARY:
Preoperative midnight NPO is a traditional method for preventing aspiration during general anesthesia. However, recent studies reported that drinking carbohydrate beverage, three hours prior the surgery helps reducing patients starving, uncomfortment, and fatigue without other complication. QOR 40 is developed for evaluating patients' recovery condition regarding physical, psychological, and social aspects. Enhanced Recovery After Surgery(ERAS) is a concept for reducing patients' hospital stay and helping recovery. Studies showed that drinking carbohydrate beverage made better recovery of bowel function and shorter hospital stay in colorectal surgeries. However, the effect of carbohydrate drink for laparoscopic surgery is not yet proved. Therefore, the investigators will show the effect of carbohydrate drinking through this study.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic colorectal surgery,
* 20~85 year-old patients

Exclusion Criteria:

* diabetes mellitus
* Inability to consume clear fluids
* GERD or gastrointestinal obstruction
* Liver cirrhosis
* corticosteroid treatment
* ASA>4
* starting surgery five and more hours after drinking carbohydrate beverage
* pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
total score of a survey using Quality of Recovery 40 | 1 day

SECONDARY OUTCOMES:
amount of perioperative water intake | 1 day
  measure with ml
amount of perioperative urine output | 1 day
  measure with ml
time to bowel function recovery | 1 day
hospital stay duration from operation to discharge | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107